CLINICAL TRIAL: NCT03824158
Title: Patient-centered and Efficacious Advance Care Planning in Cancer: the PEACe Comparative Effectiveness Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Yael Schenker, MD, MAS, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY19080337; 1R01CA235730-01 (NIH)
Record Dates: First submitted 2019-01-24; First posted 2019-01-31 (Actual); Results first posted 2025-01-17 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Cancer; Advance Care Planning
Keywords: cancer, advance care planning
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Facilitated advance care planning (in-person or telephonic) (Active Comparator): Patients randomized to this arm will participate in in-person or telephonic facilitated advance care planning (ACP) discussions using the Respecting Choices model.
  Interventions: Behavioral: Facilitated advance care planning (in-person or telephonic)
- Web-based advance care planning (Active Comparator): Patients randomized to this arm will participate in web-based ACP via the PREPARE website.
  Interventions: Behavioral: Web-based advance care planning

INTERVENTIONS:
Behavioral: Facilitated advance care planning (in-person or telephonic) — The facilitator will contact the patient to schedule the ACP discussion. ACP discussions will be led by a nurse or social worker with supportive oncology experience who has been trained as a Respecting Choices facilitator, include the patient's caregiver when available, last 45-60 minutes, and be held in a private location at or near the patient's oncology clinic, or telephonically. Facilitators will use a structured interview tool as a discussion roadmap and provide guidance in choosing a medical decision maker, exploring serious illness understanding and experiences, identifying goals and values, and making future treatment decisions. Facilitators will provide a copy of a written advance directive, assist with completion when appropriate, and make recommendations for communicating goals and sharing written preferences.
  Arms: Facilitated advance care planning (in-person or telephonic)
Behavioral: Web-based advance care planning — Instructions for accessing and using the PREPARE website will be shared with participants upon randomization. Patients and their caregivers review the 5 steps of PREPARE (approximately 10 minutes per step) and create an action plan for each step. The PREPARE website includes a link to a written advance directive that participants are able to complete. The PREPARE website can be reviewed on a home computer or on a tablet in the oncology practice.
  Arms: Web-based advance care planning

SUMMARY:
The overall goal of this study is to identify the most effective and efficient advance care planning (ACP) strategy for patients with advanced cancer.

The specific aims are to:

Aim 1. Compare the effectiveness of in-person, facilitated ACP versus web-based ACP on patient and family caregiver outcomes.

Aim 2. Assess implementation costs and the effects of in-person, facilitated ACP and web-based ACP on healthcare utilization at end of life.

Aim 3. Identify contexts and mechanisms that influence the effectiveness of in-person, facilitated ACP versus web-based ACP.

DETAILED DESCRIPTION:
Study investigators will conduct a single-blind, patient-level randomized trial to compare the effectiveness of two different patient-facing advance care planning (ACP) interventions. Investigators will enroll 400 patients with advanced cancer and their family caregivers to receive either (1) in-person discussions with trained facilitators or (2) web-based ACP using interactive videos. Because these approaches have never been compared directly, it is unclear whether one form of advance care planning is more potent, and if so, for whom and under what circumstances.

Aim 1 compares the effectiveness of in-person, facilitated ACP versus web-based ACP on patient and family caregiver outcomes (ACP engagement, ACP discussions, advance directive completion, goal attainment, and caregiver psychological symptoms). Aim 2 assesses implementation costs of each intervention and effects on healthcare utilization at end of life. Aim 3 identifies contexts and mechanisms influencing the effectiveness of each approach. Primary patient outcomes will be assessed at 12 weeks. Participants will be followed until 12 weeks after the patient's death or completion of the 48-month data collection period, whichever occurs first. In-depth interviews with patients, caregivers, and clinicians will begin in Year 2 of the grant and continue until thematic saturation is reached.

ELIGIBILITY:
Patient Inclusion Criteria:

1. 18 years of age or older
2. Solid tumor
3. The oncologist "would not be surprised" if the patient died within the next year
4. Eastern Cooperative Oncology Group performance status (ECOG PS) of 0, 1, or 2
5. Planning to receive ongoing care at a participating oncology clinic
6. Willing to participate in either a web-based or facilitated program

Patient Exclusion Criteria:

1. Does not speak English
2. Inability to consent, using a validated teach-back method
3. Hematologic malignancy
4. No phone for additional study contacts and follow-up interviews
5. Unable to participate in advance care planning, as assessed by clinician
6. Unable to complete the baseline interview

Patients will be able to identify and enroll a caregiver, designated by the patient as the primary family member or friend involved in their care and best able to participate in the study.

Caregiver Inclusion criteria:

1. 18 years of age or older
2. Family member or friend of an eligible patient
3. Primary person involved in patient's care and best able to participate in the study, as assessed by patient

Caregiver Exclusion criteria:

1. Does not speak English
2. No phone for additional study contacts and follow-up interviews
3. Unable to complete the baseline interview

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 672 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2025-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yael Schenker, MD, MPH, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schenker Y, Belin SC, Wang T, Sudore RL, Hammes B, Arnold RM, Flowers R, Chiu E, Hall J, Dudley-Morrissey Y, Ferrell B, Crowley-Matoka M, Brufsky A, Chu E, Gorantla V, Mehta D, Thomas R, Yee M, White D. Facilitated Versus Patient-Directed Advance Care Planning Among Patients With Advanced Cancer: A Randomized Clinical Trial. JCO Oncol Pract. 2025 Oct;21(10):1447-1457. doi: 10.1200/OP-25-00046. Epub 2025 Mar 19. PMID 40106743

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred from August 1, 2019 until July 14, 2023. Patients were enrolled from 8 oncology clinics within the University of Pittsburgh Medical Center Hillman Cancer Center Network in western Pennsylvania. Patients were encouraged but not required to identify a caregiver, defined as the primary adult (family member or friend) involved in their care and best able to participate in the study, as assessed by the patient. Patients without a willing caregiver participant were not excluded.
Groups:
- Web-based Advance Care Planning (PATIENTS): Patients randomized to this arm will participate in web-based ACP via the PREPARE website.
  Web-based advance care planning: Instructions for accessing and using the PREPARE website will be shared with participants upon randomization. Patients and their caregivers review the 5 steps of PREPARE (approximately 10 minutes per step) and create an action plan for each step. The PREPARE website includes a link to a written advance directive that participants are able to complete. The PREPARE website can be reviewed on a home computer or on a tablet in the oncology practice.
- Facilitated Advance Care Planning (In-person or Telephonic) (PATIENTS): Patients randomized to this arm will participate in in-person or telephonic facilitated advance care planning (ACP) discussions using the Respecting Choices model.
  Facilitated advance care planning (in-person or telephonic): The facilitator will contact the patient to schedule the ACP discussion. ACP discussions will be led by a nurse or social worker with supportive oncology experience who has been trained as a Respecting Choices facilitator, include the patient's caregiver when available, last 45-60 minutes, and be held in a private location at or near the patient's oncology clinic, or telephonically. Facilitators will use a structured interview tool as a discussion roadmap and provide guidance in choosing a medical decision maker, exploring serious illness understanding and experiences, identifying goals and values, and making future treatment decisions. Facilitators will provide a copy of a written advance directive, assist with completion when appropriate, and make recommendations for communicating goals and sharing written preferences.
- Web-based Advance Care Planning (CAREGIVERS): Enrolled caregivers of patients randomized to the web-based advance care planning arm.
- Facilitated Advance Care Planning (In-person or Telephonic) (CAREGIVERS): Enrolled caregivers of patients randomized to the facilitated advance care planning arm.
Period: Overall Study
Arm/Group | Web-based Advance Care Planning (PATIENTS) | Facilitated Advance Care Planning (In-person or Telephonic) (PATIENTS) | Web-based Advance Care Planning (CAREGIVERS) | Facilitated Advance Care Planning (In-person or Telephonic) (CAREGIVERS)
Started | 203 | 197 | 133 | 139
Completed | 134 | 135 | 102 | 108
Not Completed | 69 | 62 | 31 | 31

BASELINE CHARACTERISTICS:
Population: Some baseline measures were only collected for either patients or caregivers.
Groups:
- Total: Total of all reporting groups
Arm/Group | Web-based Advance Care Planning (PATIENTS) | Facilitated Advance Care Planning (In-person or Telephonic) (PATIENTS) | Web-based Advance Care Planning (CAREGIVERS) | Facilitated Advance Care Planning (In-person or Telephonic) (CAREGIVERS) | Total
Number analyzed (Participants) | 203 | 197 | 133 | 139 | 672
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.8 (10) | 68.1 (11) | 62.2 (13.6) | 61.9 (13.5) | 67.9 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 96 | 96 | 103 | 391
  Male | 107 | 101 | 37 | 36 | 281
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 1 | 1 | 6
  Not Hispanic or Latino | 201 | 194 | 132 | 136 | 663
  Unknown or Not Reported | 1 | 0 | 0 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1 | 2
  Asian | 1 | 1 | 1 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 17 | 13 | 6 | 5 | 41
  White | 184 | 181 | 125 | 132 | 622
  More than one race | 1 | 1 | 1 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 203 | 197 | 133 | 139 | 672
Education Level [Count of Participants; unit: Participants] — Participants self-reported their highest level of formal education completed at the time of enrollment.
  Participants
    < High school | 4 | 6 | 1 | 3 | 14
    High school diploma or GED | 66 | 63 | 34 | 36 | 199
    Some college or college degree | 107 | 99 | 74 | 69 | 349
    Graduate or professional degree | 25 | 28 | 24 | 31 | 108
    Refused to answer | 1 | 1 | 0 | 0 | 2
Current Marital Status [Count of Participants; unit: Participants] — Participants self-reported their current marital status at the time of enrollment.
  Participants
    Never married | 16 | 14 | 12 | 6 | 48
    Married | 125 | 118 | 105 | 113 | 461
    Widowed | 28 | 35 | 6 | 9 | 78
    Divorced/Separated | 28 | 28 | 8 | 10 | 74
    Refused to answer | 5 | 0 | 2 | 1 | 8
    Unknown | 1 | 2 | 0 | 0 | 3
Ability to manage on income [Count of Participants; unit: Participants] — Participants self-reported their ability to manage on their income at the time of enrollment.
  Participants
    Cannot make ends meet | 6 | 2 | 8 | 2 | 18
    Just manage to get by | 51 | 46 | 21 | 24 | 142
    Have enough with a little extra | 59 | 77 | 58 | 54 | 248
    Money is not a problem | 56 | 48 | 35 | 41 | 180
    Refused to answer | 27 | 24 | 11 | 18 | 80
    Unknown | 4 | 0 | 0 | 0 | 4
Religion [Count of Participants; unit: Participants] — Participants self-reported their religion at the time of enrollment.
  Participants
    Agnostic/Atheist/No religion | 8 | 14 | 5 | 9 | 36
    Buddhist | 1 | 0 | 0 | 0 | 1
    Catholic | 91 | 72 | 57 | 56 | 276
    Other Christian | 24 | 27 | 12 | 19 | 82
    Hindu | 0 | 1 | 0 | 1 | 2
    Jewish | 3 | 5 | 3 | 4 | 15
    Muslim | 0 | 0 | 1 | 0 | 1
    Protestant | 42 | 48 | 33 | 28 | 151
    Declined to answer | 18 | 16 | 9 | 8 | 51
    Other | 15 | 14 | 13 | 14 | 56
    Unknown | 1 | 0 | 0 | 0 | 1
Religious importance [Count of Participants; unit: Participants] — Participants self-reported how important religion is to them at the time of enrollment.
  Participants
    Not at all important | 9 | 20 | 2 | 8 | 39
    Not too important | 24 | 25 | 17 | 21 | 87
    Fairly important | 53 | 43 | 39 | 43 | 178
    Very important | 106 | 101 | 68 | 64 | 339
    Refused to answer | 10 | 7 | 7 | 3 | 27
    Unknown | 1 | 1 | 0 | 0 | 2
Confidence filling out medical forms [Count of Participants; unit: Participants] — Participants self-reported how confident they are filling out medical forms at the time of enrollment.
  Participants
    Not at all | 6 | 7 | 1 | 3 | 17
    A little bit | 9 | 9 | 4 | 3 | 25
    Somewhat | 54 | 43 | 16 | 15 | 128
    Quite a bit | 40 | 47 | 31 | 33 | 151
    Extremely | 94 | 91 | 81 | 85 | 351
How many other people live in your household? [Count of Participants; unit: Participants] — Participants self-reported how many other people currently live in their household at the time of enrollment.
  Participants
    0 | 45 | 49 | 7 | 10 | 111
    1 | 112 | 110 | 90 | 95 | 407
    2 | 26 | 24 | 17 | 17 | 84
    3 | 14 | 12 | 14 | 14 | 54
    4+ | 4 | 1 | 5 | 3 | 13
    Unknown | 2 | 1 | 0 | 0 | 3
Current employment status [Count of Participants; unit: Participants] — Participants self-reported their current employment status at the time of enrollment.
  Participants
    Working full-time | 20 | 21 | 40 | 46 | 127
    Working part-time | 7 | 7 | 11 | 12 | 37
    Unemployed | 11 | 9 | 3 | 2 | 25
    Retired | 118 | 120 | 59 | 62 | 359
    Homemaker (never worked for pay) | 1 | 4 | 5 | 3 | 13
    Disability | 24 | 22 | 4 | 6 | 56
    Other | 16 | 11 | 10 | 7 | 44
    Refused to answer | 6 | 3 | 1 | 1 | 11
HADS Survey Depression Subscale Scores [Mean (Standard Deviation); unit: score on a scale] — The Hospital Anxiety and Depression Scale (HADS) is a 14-item scale designed to measure anxiety and depression. Subscale scores range 0-21, with higher scores indicating higher anxiety or depression.
  score on a scale | 4.62 (3.44) | 4.69 (3.52) | 4.22 (3.54) | 3.96 (3.43) | 4.65 (3.48)
HADS Survey Anxiety Subscale Scores [Mean (Standard Deviation); unit: score on a scale] — The Hospital Anxiety and Depression Scale (HADS) is a 14-item scale designed to measure anxiety and depression. Subscale scores range 0-21, with higher scores indicating higher anxiety or depression.
  score on a scale | 5.22 (3.69) | 5.15 (3.73) | 7.0 (4.1) | 7.44 (4.43) | 5.19 (3.71)
Current living situation [Count of Participants; unit: Participants] — Participants self-reported their current living situation at the time of enrollment. Population: Current living situation was only collected for enrolled patients. Caregivers were not included in this measure.
  Participants
    number analyzed (Participants) | 203 | 197 | 0 | 0 | 400
    In a home I (or my family) own | 161 | 155 |  |  | 316
    In a home I (or my family) rent | 31 | 28 |  |  | 59
    In a Board and Care home | 0 | 0 |  |  | 0
    In an Assisted Living Facility | 2 | 3 |  |  | 5
    In a Nursing Home | 0 | 3 |  |  | 3
    Other/Unsure | 6 | 8 |  |  | 14
    Refused to answer | 3 | 0 |  |  | 3
Cancer type [Count of Participants; unit: Participants] — Cancer type was collected at the time of enrollment by patient self-report, followed by querying the oncologist and/or checking the medical record to confirm accuracy of the self-reported cancer type. Population: Cancer type was only collected for enrolled patients. Caregivers were not included in this measure.
  Participants
    number analyzed (Participants) | 203 | 197 | 0 | 0 | 400
    Genitourinary | 21 | 20 |  |  | 41
    Brain | 1 | 0 |  |  | 1
    Breast | 18 | 31 |  |  | 49
    Gynecologic | 7 | 12 |  |  | 19
    Gastrointestinal | 39 | 38 |  |  | 77
    Hepatobiliary | 9 | 8 |  |  | 17
    Head and Neck | 10 | 10 |  |  | 20
    Lung | 48 | 34 |  |  | 82
    Melanoma | 1 | 0 |  |  | 1
    Pancreatic | 20 | 22 |  |  | 42
    Prostate | 23 | 18 |  |  | 41
    Other | 6 | 4 |  |  | 10
Time since first diagnosed with cancer [Count of Participants; unit: Participants] — Patients self-reported the amount of time since they were first diagnosed with cancer. Population: Time since first diagnosed with cancer was only collected for enrolled patients. Caregivers were not included in this measure.
  Participants
    number analyzed (Participants) | 203 | 197 | 0 | 0 | 400
    Less than one month ago | 11 | 6 |  |  | 17
    ≥ 1 month but < 6 months ago | 27 | 31 |  |  | 58
    ≥ 6 months but < 1 year ago | 44 | 43 |  |  | 87
    ≥ 1 year but < 2 years ago | 31 | 23 |  |  | 54
    ≥ 2 years but < 5 years ago | 36 | 39 |  |  | 75
    ≥ 5 years ago | 49 | 53 |  |  | 102
    Refused to answer | 4 | 2 |  |  | 6
    Unknown | 1 | 0 |  |  | 1
Time receiving care from current oncologist [Count of Participants; unit: Participants] — Patients self-reported the amount of time they have been receiving care from their current oncologist. Population: Time receiving care from current oncologist was only collected for enrolled patients. Caregivers were not included in this measure.
  Participants
    number analyzed (Participants) | 203 | 197 | 0 | 0 | 400
    Less than one month | 13 | 11 |  |  | 24
    ≥ 1 month but < 6 months | 40 | 36 |  |  | 76
    ≥ 6 months but < 1 year | 48 | 51 |  |  | 99
    ≥ 1 year but < 2 years | 35 | 29 |  |  | 64
    ≥ 2 years but < 5 years | 41 | 39 |  |  | 80
    ≥ 5 years | 23 | 31 |  |  | 54
    Refused to answer | 3 | 0 |  |  | 3
ECOG Performance Status [Count of Participants; unit: Participants] — The Eastern Cooperative Oncology Group (ECOG) Performance Status scale describes how well cancer patients can function in daily life. Scores range 0-5; higher scores indicate greater functional impairment. Scores were collected for the study by querying treating oncologist. 0=Fully active, able to carry on all pre-disease performance w/o restriction 1=Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature 2=Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours. Population: ECOG score was only collected for enrolled patients. Caregivers were not included in this measure.
  Participants
    number analyzed (Participants) | 203 | 197 | 0 | 0 | 400
    ECOG Score - 0 | 64 | 68 |  |  | 132
    ECOG Score - 1 | 122 | 102 |  |  | 224
    ECOG Score - 2 | 17 | 27 |  |  | 44
Patient reported previously completing a living will or advance directive [Count of Participants; unit: Participants] — Binary question, YES or NO, with YES indicating the patient reported previously completed a living will or advance directive. Population: Previous living will or advance directive completion was only collected for enrolled patients. Caregivers were not included in this measure.
  Participants
    number analyzed (Participants) | 203 | 197 | 0 | 0 | 400
    (all) | 95 | 103 |  |  | 198
Patient reported previously having advance care planning discussions with caregivers [Count of Participants; unit: Participants] — Binary question, YES or NO, with YES indicating the patient reported previously having advance care planning discussions with caregivers. Population: Previous advance care planning discussions were only collected for enrolled patients. Caregivers were not included in this measure.
  Participants
    number analyzed (Participants) | 203 | 197 | 0 | 0 | 400
    (all) | 139 | 136 |  |  | 275
Patient reported previously having advance care planning discussions with physicians [Count of Participants; unit: Participants] — Binary question, YES or NO, with YES indicating the patient reported previously having advance care planning discussions with physicians. Population: Previous advance care planning discussions were only collected for enrolled patients. Caregivers were not included in this measure.
  Participants
    number analyzed (Participants) | 203 | 197 | 0 | 0 | 400
    (all) | 48 | 53 |  |  | 101
Prior living will or advance directive in the medical record [Count of Participants; unit: Participants] — The patient's electronic medical record was reviewed to determine if a living will or advance directive was uploaded and available to view prior to the study intervention. Population: Living will or advance directive information was collected only for patients.
  Participants
    number analyzed (Participants) | 203 | 197 | 0 | 0 | 400
    (all) | 24 | 27 |  |  | 51
Prior POLST form in the medical record [Count of Participants; unit: Participants] — The patient's electronic medical record was reviewed to determine if a Physician Orders for Life-Sustaining Treatment (POLST) form was uploaded and available to view prior to the study intervention. Population: POLST form information was collected only for patients.
  Participants
    number analyzed (Participants) | 203 | 197 | 0 | 0 | 400
    (all) | 4 | 8 |  |  | 12
Advance Care Planning (ACP) Engagement Survey Total Scores [Mean (Standard Deviation); unit: score on a scale] — 15-item Advance Care Planning (ACP) engagement survey assesses ACP processes related to choosing a medical decision maker, discussing and documenting preference for care at end of life, flexibility for surrogate decision making, and asking questions of medical providers. A single summary score will be reported (range 0-5 with higher scores indicating higher engagement). Population: Advance Care Planning Engagement scores were only collected for enrolled patients. Caregivers were not included in this measure.
  score on a scale
    number analyzed (Participants) | 203 | 197 | 0 | 0 | 400
    (all) | 3.66 (0.93) | 3.74 (1.02) |  |  | 3.70 (0.98)
Relationship to enrolled patient [Count of Participants; unit: Participants] — Caregivers self-reported their relationship to the enrolled patient at the time of enrollment. Population: Relationship to enrolled patient was only collected for caregivers.
  Participants
    number analyzed (Participants) | 0 | 0 | 133 | 139 | 272
    Spouse/partner |  |  | 90 | 85 | 175
    Child |  |  | 25 | 24 | 49
    Parent |  |  | 5 | 4 | 9
    Sibling |  |  | 6 | 12 | 18
    Friend |  |  | 2 | 5 | 7
    Other |  |  | 4 | 9 | 13
    Refused to answer |  |  | 1 | 0 | 1
Caregiver lives with the patient [Count of Participants; unit: Participants] — Binary question, YES or NO, with YES indicating the caregiver reported living with the patient at the time of enrollment. Population: Living with the enrolled patient was only collected for caregivers.
  Participants
    number analyzed (Participants) | 0 | 0 | 133 | 139 | 272
    (all) |  |  | 98 | 94 | 192
Current care provider for the patient [Count of Participants; unit: Participants] — Binary question, YES or NO, with YES indicating the caregiver reported being a current care provider for the patient at the time of enrollment. Population: Care provider status was only collected for caregivers.
  Participants
    number analyzed (Participants) | 0 | 0 | 133 | 139 | 272
    (all) |  |  | 117 | 124 | 241
Average days per week providing care [Mean (Standard Deviation); unit: days per week] — Caregivers self-reported the average number of days per week they provide care to the patient. Population: Average days providing care was only collected for caregivers.
  days per week
    number analyzed (Participants) | 0 | 0 | 133 | 139 | 272
    (all) |  |  | 5.33 (2.3) | 5.59 (2.3) | 5.46 (2.3)
Average hours per day providing care [Mean (Standard Deviation); unit: hours per day] — Caregivers self-reported the average number of hours per day they provide care to the patient. Population: Average hours providing care was only collected for caregivers.
  hours per day
    number analyzed (Participants) | 0 | 0 | 133 | 139 | 272
    (all) |  |  | 6.92 (8.1) | 7.15 (7.9) | 7.03 (8.0)
Currently providing care for anyone else [Count of Participants; unit: Participants] — Caregivers self-reported if they are currently providing care for anyone other than the enrolled patient. Population: Providing care for anyone else was only collected for caregivers.
  Participants
    number analyzed (Participants) | 0 | 0 | 133 | 139 | 272
    (all) |  |  | 29 | 31 | 60

OUTCOME MEASURES:

1. Primary Outcome: Advance Care Planning Engagement
Description: 15-item Advance Care Planning (ACP) engagement survey assesses ACP processes related to choosing a medical decision maker, discussing and documenting preference for care at end of life, flexibility for surrogate decision making, and asking questions of medical providers. A single summary score will be reported (range 0-5 with higher scores indicating higher engagement).
Time Frame: 12 weeks
Population: Number of participants that completed 12 week outcomes assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Web-based Advance Care Planning (PATIENTS) | Facilitated Advance Care Planning (In-person or Telephonic) (PATIENTS)
Number analyzed (Participants) | 134 | 135
score on a scale | 4.08 (0.82) | 4.34 (0.78)
Statistical Analysis 1: Comparison: Web-based Advance Care Planning (PATIENTS) vs Facilitated Advance Care Planning (In-person or Telephonic) (PATIENTS); Test type: Superiority; p = 0.0014, Mixed Models Analysis

2. Secondary Outcome: Number of Participants Who Have Had Advance Care Planning Discussions With Caregivers
Description: "Has [participant] talked with [participant's] family or friends about the kind of medical care [participant] would want if [participant] were very sick or near the end of life?"
Time Frame: 12 weeks
Population: Number of participants that completed 12 week outcomes assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Web-based Advance Care Planning (PATIENTS) | Facilitated Advance Care Planning (In-person or Telephonic) (PATIENTS)
Number analyzed (Participants) | 134 | 135
Participants | 117 | 120
Statistical Analysis 1: Comparison: Web-based Advance Care Planning (PATIENTS) vs Facilitated Advance Care Planning (In-person or Telephonic) (PATIENTS); Test type: Superiority; p = 0.76, Regression, Logistic

3. Secondary Outcome: Number of Participants Who Have Had Advance Care Planning Discussions With Physicians
Description: "Has [participant] talked with [participant's] doctor about the kind of medical care [participant] would want if [participant] were very sick or near the end of life?"
Time Frame: 12 weeks
Population: Number of participants that completed 12 week outcomes assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Web-based Advance Care Planning (PATIENTS) | Facilitated Advance Care Planning (In-person or Telephonic) (PATIENTS)
Number analyzed (Participants) | 134 | 135
Participants | 54 | 67
Statistical Analysis 1: Comparison: Web-based Advance Care Planning (PATIENTS) vs Facilitated Advance Care Planning (In-person or Telephonic) (PATIENTS); Test type: Superiority; p = 0.13, Mixed Models Analysis

4. Secondary Outcome: Number of Participants Who Have Completed an Advance Directive
Description: "Has [participant] completed a living will or advance directive?"
Time Frame: 12 weeks
Population: Number of participants that completed 12 week outcomes assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Web-based Advance Care Planning (PATIENTS) | Facilitated Advance Care Planning (In-person or Telephonic) (PATIENTS)
Number analyzed (Participants) | 134 | 135
Participants | 80 | 101
Statistical Analysis 1: Comparison: Web-based Advance Care Planning (PATIENTS) vs Facilitated Advance Care Planning (In-person or Telephonic) (PATIENTS); Test type: Superiority; p = 0.008, Mixed Models Analysis

5. Secondary Outcome: Documented Care Goals
Description: Investigators will assess documented care goals by reviewing medical records for any care goals documented since baseline (Yes/No).
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | Web-based Advance Care Planning (PATIENTS) | Facilitated Advance Care Planning (In-person or Telephonic) (PATIENTS)
Number analyzed (Participants) | 203 | 197
participants
  New advance directive or living will | 4 | 18
  New Physician Orders for Life-sustaining Treatment (POLST) form | 1 | 8
  New Code Status | 29 | 31
  New Goals of Care discussion | 26 | 22
Statistical Analysis 1: Comparison: Web-based Advance Care Planning (PATIENTS) vs Facilitated Advance Care Planning (In-person or Telephonic) (PATIENTS); Advance directive or living will; Test type: Superiority; p = 0.002, Chi-squared
Statistical Analysis 2: Comparison: Web-based Advance Care Planning (PATIENTS) vs Facilitated Advance Care Planning (In-person or Telephonic) (PATIENTS); POLST; Test type: Superiority; p = 0.02, Fisher Exact
Statistical Analysis 3: Comparison: Web-based Advance Care Planning (PATIENTS) vs Facilitated Advance Care Planning (In-person or Telephonic) (PATIENTS); Code Status; Test type: Superiority; p = 0.78, Chi-squared
Statistical Analysis 4: Comparison: Web-based Advance Care Planning (PATIENTS) vs Facilitated Advance Care Planning (In-person or Telephonic) (PATIENTS); Goals of Care discussion; Test type: Superiority; p = 0.61, Chi-squared

6. Secondary Outcome: Caregiver Depression Symptoms
Description: Depression subscale of the 14-item Hospital Anxiety and Depression Scale (HADS) will be used to assess caregiver depression symptoms at 12 weeks and bereavement. The HADS depression subscale scores range from 0 to 21, with higher scores indicating more distress.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Web-based Advance Care Planning (CAREGIVERS) | Facilitated Advance Care Planning (In-person or Telephonic) (CAREGIVERS)
Number analyzed (Participants) | 102 | 108
score on a scale | 4.34 (4.07) | 3.69 (3.57)
Statistical Analysis 1: Comparison: Web-based Advance Care Planning (CAREGIVERS) vs Facilitated Advance Care Planning (In-person or Telephonic) (CAREGIVERS); Test type: Superiority; p = 0.17, Mixed Models Analysis

7. Secondary Outcome: Caregiver Anxiety Symptoms
Description: Anxiety subscale of the 14-item Hospital Anxiety and Depression Scale (HADS) will be used to assess caregiver anxiety symptoms at 12 weeks and bereavement. The anxiety subscale scores range from 0 to 21, with higher scores indicating more distress.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Web-based Advance Care Planning (CAREGIVERS) | Facilitated Advance Care Planning (In-person or Telephonic) (CAREGIVERS)
Number analyzed (Participants) | 102 | 108
score on a scale | 6.94 (4.6) | 6.5 (3.92)
Statistical Analysis 1: Comparison: Web-based Advance Care Planning (CAREGIVERS) vs Facilitated Advance Care Planning (In-person or Telephonic) (CAREGIVERS); Test type: Superiority; p = 0.11, Mixed Models Analysis

8. Secondary Outcome: Receipt of Goal-concordant End-of-life Care - Patient Wishes Followed
Description: Bereaved caregivers will be asked "In [participant's] opinion, to what extent were [the patient's] wishes followed in the medical care received in the last month of life?" Receipt of goal-concordant end-of-life care - patient wishes followed will be defined as care that "followed patients' wishes a great deal."
Time Frame: during bereavement, up to 60 months
Population: Bereaved caregivers
Measure: Count of Participants; unit: Participants
Arm/Group | Web-based Advance Care Planning (CAREGIVERS) | Facilitated Advance Care Planning (In-person or Telephonic) (CAREGIVERS)
Number analyzed (Participants) | 50 | 48
Participants
  A great deal | 37 | 46
  Somewhat | 11 | 2
  Not at all | 1 | 0
  Did not answer | 1 | 0
Statistical Analysis 1: Comparison: Web-based Advance Care Planning (CAREGIVERS) vs Facilitated Advance Care Planning (In-person or Telephonic) (CAREGIVERS); Test type: Superiority; p = 0.01, Fisher Exact

9. Secondary Outcome: Receipt of Goal-concordant End-of-life Care - Place of Death
Description: Bereaved caregivers will be asked about patient's preferred and actual places of death, with questions separated in the survey to minimize conscious comparison. Receipt of goal-concordant end-of-life care - place of death will be defined as patients dying in their preferred location.
Time Frame: during bereavement, up to 60 months
Population: Bereaved caregivers
Measure: Count of Participants; unit: Participants
Arm/Group | Web-based Advance Care Planning (CAREGIVERS) | Facilitated Advance Care Planning (In-person or Telephonic) (CAREGIVERS)
Number analyzed (Participants) | 50 | 48
Participants | 34 | 37
Statistical Analysis 1: Comparison: Web-based Advance Care Planning (CAREGIVERS) vs Facilitated Advance Care Planning (In-person or Telephonic) (CAREGIVERS); Test type: Superiority; p = 0.83, Fisher Exact

10. Secondary Outcome: Quality of End-of-life Care
Description: 13-item Caregiver Evaluation of Quality of End-of-Life Care (CEQUEL) scale. Total score range is 13-26, with higher scores indicating better perceived quality of care. Prolongation of Death, Perceived Suffering, and Preparation for the Death Subscales range 3-6, with higher scores indicating a better outcome. Shared Decision-Making subscale range is 4-8, with higher scores indicating a better outcome.
Time Frame: during bereavement, up to 60 months
Population: Bereaved caregivers
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Web-based Advance Care Planning (CAREGIVERS) | Facilitated Advance Care Planning (In-person or Telephonic) (CAREGIVERS)
Number analyzed (Participants) | 50 | 48
score on a scale
  Prolongation of Death subscale | 5.62 (0.78) | 5.69 (0.62)
  Perceived Suffering Subscale | 5.51 (0.83) | 5.45 (0.91)
  Shared Decision-Making subscale | 7.67 (0.74) | 7.7 (0.68)
  Preparation for the Death subscale | 5.66 (0.72) | 5.51 (0.72)
  Total Score | 24.45 (2.05) | 24.35 (1.83)
Statistical Analysis 1: Comparison: Web-based Advance Care Planning (CAREGIVERS) vs Facilitated Advance Care Planning (In-person or Telephonic) (CAREGIVERS); Test type: Superiority; p = 0.32, Wilcoxon (Mann-Whitney) — Total Score p-value

11. Secondary Outcome: Caregiver Post-traumatic Stress Symptoms
Description: 22-item Impact of Events Scale-revised has a scoring range from 0-88, with a higher total score indicating more post-traumatic stress symptoms. Avoidance, Intrusions, and Hyperarousal Subscales range 0-4, with higher scores indicating a worse outcome.
Time Frame: during bereavement, up to 60 months
Population: Bereaved caregivers
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Web-based Advance Care Planning (CAREGIVERS) | Facilitated Advance Care Planning (In-person or Telephonic) (CAREGIVERS)
Number analyzed (Participants) | 50 | 48
score on a scale
  Avoidance subscale | 1.15 (0.64) | 0.96 (0.79)
  Intrusions Subscale | 1.99 (0.89) | 1.48 (0.86)
  Hyperarousal Subscale | 1.06 (0.84) | 0.74 (0.64)
  IES-R Total Score | 31.5 (15.2) | 23.9 (14.6)
Statistical Analysis 1: Comparison: Web-based Advance Care Planning (CAREGIVERS) vs Facilitated Advance Care Planning (In-person or Telephonic) (CAREGIVERS); IES-R Total Score p-value; Test type: Superiority; p = 0.01, t-test, 2 sided

12. Secondary Outcome: Caregiver Depression Symptoms
Description: as for outcome 6
Time Frame: bereavement, up to 60 months
Population: Bereaved caregivers
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Web-based Advance Care Planning (CAREGIVERS) | Facilitated Advance Care Planning (In-person or Telephonic) (CAREGIVERS)
Number analyzed (Participants) | 50 | 48
score on a scale | 5.87 (4.11) | 5.34 (6.56)
Statistical Analysis 1: Comparison: Web-based Advance Care Planning (CAREGIVERS) vs Facilitated Advance Care Planning (In-person or Telephonic) (CAREGIVERS); Test type: Superiority; p = 0.50, t-test, 2 sided

13. Secondary Outcome: Caregiver Anxiety Symptoms
Description: as for outcome 7
Time Frame: during bereavement, up to 60 months
Population: Bereaved caregivers
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Web-based Advance Care Planning (CAREGIVERS) | Facilitated Advance Care Planning (In-person or Telephonic) (CAREGIVERS)
Number analyzed (Participants) | 50 | 48
score on a scale | 6.72 (4.59) | 6.56 (3.32)
Statistical Analysis 1: Comparison: Web-based Advance Care Planning (CAREGIVERS) vs Facilitated Advance Care Planning (In-person or Telephonic) (CAREGIVERS); Test type: Superiority; p = 0.84, t-test, 2 sided

14. Other Pre Specified Outcome: Number of Participants Who Received Chemotherapy Within Last 2 Weeks of Life
Description: Investigators will measure whether chemotherapy was administered within the last 2 weeks of life (Y/N)
Time Frame: Assessed after patient death
Population: Deceased patients
Measure: Count of Participants; unit: Participants
Arm/Group | Web-based Advance Care Planning (PATIENTS) | Facilitated Advance Care Planning (In-person or Telephonic) (PATIENTS)
Number analyzed (Participants) | 112 | 116
Participants | 12 | 5
Statistical Analysis 1: Comparison: Web-based Advance Care Planning (PATIENTS) vs Facilitated Advance Care Planning (In-person or Telephonic) (PATIENTS); Test type: Superiority; p = 0.07, Chi-squared

15. Other Pre Specified Outcome: Number of Participants Admitted to an Intensive Care Unit Within Last 30 Days of Life
Description: Investigators will measure whether participant was admitted to the intensive care unit in the last 30 days of life (Y/N)
Time Frame: Assessed after patient death
Population: Deceased patients
Measure: Count of Participants; unit: Participants
Arm/Group | Web-based Advance Care Planning (PATIENTS) | Facilitated Advance Care Planning (In-person or Telephonic) (PATIENTS)
Number analyzed (Participants) | 112 | 116
Participants | 20 | 16
Statistical Analysis 1: Comparison: Web-based Advance Care Planning (PATIENTS) vs Facilitated Advance Care Planning (In-person or Telephonic) (PATIENTS); Test type: Superiority; p = 0.4, Chi-squared

16. Other Pre Specified Outcome: Number of Participants Admitted to Hospice Within Last 30 Days of Life
Description: Investigators will measure whether the participant was admitted to hospice (Y/N)
Time Frame: Assessed after patient death
Population: Deceased patients
Measure: Count of Participants; unit: Participants
Arm/Group | Web-based Advance Care Planning (PATIENTS) | Facilitated Advance Care Planning (In-person or Telephonic) (PATIENTS)
Number analyzed (Participants) | 112 | 116
Participants | 64 | 76
Statistical Analysis 1: Comparison: Web-based Advance Care Planning (PATIENTS) vs Facilitated Advance Care Planning (In-person or Telephonic) (PATIENTS); Test type: Superiority; p = 0.19, Chi-squared

17. Other Pre Specified Outcome: Number of Participants Admitted to Hospice Within Last 3 Days of Life
Description: Investigators will measure whether the participant was admitted to hospice for < 3 days (Y/N)
Time Frame: Assessed after patient death
Population: Deceased patients
Measure: Count of Participants; unit: Participants
Arm/Group | Web-based Advance Care Planning (PATIENTS) | Facilitated Advance Care Planning (In-person or Telephonic) (PATIENTS)
Number analyzed (Participants) | 112 | 116
Participants | 19 | 25
Statistical Analysis 1: Comparison: Web-based Advance Care Planning (PATIENTS) vs Facilitated Advance Care Planning (In-person or Telephonic) (PATIENTS); Test type: Superiority; p = 0.38, Chi-squared

18. Other Pre Specified Outcome: Healthcare Utilization at End of Life - Hospice Length of Stay
Description: For participants admitted to hospice, investigators will measure number of days in hospice.
Time Frame: Assessed after patient death
Population: Deceased patients
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Web-based Advance Care Planning (PATIENTS) | Facilitated Advance Care Planning (In-person or Telephonic) (PATIENTS)
Number analyzed (Participants) | 64 | 76
days | 15.8 (19.7) | 27.8 (41.8)
Statistical Analysis 1: Comparison: Web-based Advance Care Planning (PATIENTS) vs Facilitated Advance Care Planning (In-person or Telephonic) (PATIENTS); Test type: Superiority; p = 0.09, Wilcoxon (Mann-Whitney)

19. Other Pre Specified Outcome: Number of Participants Who Were Hospitalized Within Last 30 Days of Life
Description: Investigators will measure the number of participants hospitalized within in the last 30 days of life
Time Frame: Assess after patient death
Population: Deceased patients
Measure: Count of Participants; unit: Participants
Arm/Group | Web-based Advance Care Planning (PATIENTS) | Facilitated Advance Care Planning (In-person or Telephonic) (PATIENTS)
Number analyzed (Participants) | 112 | 116
Participants | 74 | 67
Statistical Analysis 1: Comparison: Web-based Advance Care Planning (PATIENTS) vs Facilitated Advance Care Planning (In-person or Telephonic) (PATIENTS); Test type: Superiority; p = 0.20, Chi-squared

20. Other Pre Specified Outcome: Number of Participants Who Had Emergency Department Visits Within Last 30 Days of Life
Description: Investigators will measure number of emergency department visits in the last 30 days of life
Time Frame: Assessed after patient death
Population: Deceased patients
Measure: Count of Participants; unit: Participants
Arm/Group | Web-based Advance Care Planning (PATIENTS) | Facilitated Advance Care Planning (In-person or Telephonic) (PATIENTS)
Number analyzed (Participants) | 112 | 116
Participants | 64 | 58
Statistical Analysis 1: Comparison: Web-based Advance Care Planning (PATIENTS) vs Facilitated Advance Care Planning (In-person or Telephonic) (PATIENTS); Test type: Superiority; p = 0.28, Chi-squared

21. Other Pre Specified Outcome: Advance Care Planning Implementation Costs
Description: Investigators will assess advance care planning implementation costs by tracking staff time spent on each intervention arm. Staff time costs for each intervention will be estimated by multiplying staff training and patient care time related to the intervention in hours by the average hourly wage for US nursing and social work staff of comparable levels.
Time Frame: through study completion, up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: up to 60 months
Arm/Group | Web-based Advance Care Planning (PATIENTS) | Facilitated Advance Care Planning (In-person or Telephonic) (PATIENTS) | Web-based Advance Care Planning (CAREGIVERS) | Facilitated Advance Care Planning (In-person or Telephonic) (CAREGIVERS)
All-Cause Mortality (participants affected / at risk) | 112/203 | 116/197 | 0/133 | 0/139
Serious Adverse Events (participants affected / at risk) | 0/203 | 0/197 | 0/133 | 0/139
Other Adverse Events (participants affected / at risk) | 0/203 | 1/197 | 0/133 | 0/139
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Web-based Advance Care Planning (PATIENTS) (N=203) | Facilitated Advance Care Planning (In-person or Telephonic) (PATIENTS) (N=197) | Web-based Advance Care Planning (CAREGIVERS) (N=133) | Facilitated Advance Care Planning (In-person or Telephonic) (CAREGIVERS) (N=139)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — During conversation during a non-study visit, the patient expressed suicidal ideation, and appeared distraught. Referred to psych services by the clinical team, and offered the Resolve Crisis number. Event not considered related to the study.
Homicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — During conversation during a non-study visit, the patient expressed homicidal ideation, and appeared distraught. Referred to psych services by the clinical team, and offered the Resolve Crisis number. Event not considered related to the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-17): https://cdn.clinicaltrials.gov/large-docs/58/NCT03824158/Prot_SAP_000.pdf